CLINICAL TRIAL: NCT00394589
Title: Randomised Controlled Trial Evaluating Strategies to Optimize Disease Activity Control in RA Patients Treated With Infliximab in Clinical Practice.
Brief Title: Re³ (Re-Cube: Retain Remicade® Response)(Study P04249AM3)
Acronym: Re³
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study enrollment was stopped due to insufficient subject accrual.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Integrated Therapeutics Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P04249
Record Dates: First submitted 2006-10-31; First posted 2006-11-01 (Estimated); Results first posted 2010-01-21 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Increased Frequency (Experimental): Continuing the same dose of 3 mg/kg infliximab, but at every 6 weeks
  Interventions: Drug: Infliximab Increased Frequency
- Increased Dose (Experimental): 3 mg/kg infliximab + 1 extra vial (100 mg) infliximab, every 8 weeks
  Interventions: Drug: Infliximab Increased Dose
- Control (Active Comparator): Continuation of infliximab 3 mg/kg every 8 weeks
  Interventions: Drug: Infliximab Control

INTERVENTIONS:
Drug: Infliximab Increased Frequency — Continuing the same dose of 3 mg/kg infliximab, but at every 6 weeks for 24 weeks
  Other Names: Increased Frequency
  Arms: Increased Frequency
Drug: Infliximab Increased Dose — 3 mg/kg infliximab + 1 extra vial (100 mg) infliximab every 8 weeks for 24 weeks
  Other Names: Increased Dose
  Arms: Increased Dose
Drug: Infliximab Control — Continuation of infliximab 3 mg/kg every 8 weeks for 24 weeks
  Other Names: Control
  Arms: Control

SUMMARY:
This Phase IIIb, randomized, multi-national, multi-center, blinded study of Infliximab (IFX) in subjects aged 18 and older with active RA is being conducted to assess whether increasing either the infusion dose or infusion frequency in patients presenting with a disease flare after an initial response to infliximab results in a significant improvement in disease activity.

Subjects responding to an initial infliximab treatment regimen, who flare during continuation of treatment at 3 mg/kg administered every 8 weeks, will be randomly assigned to one of 3 different dosing regimens of infliximab and will be treated for 4 or 5 consecutive infusions for a total duration of 24 weeks. The infliximab control group and the infliximab increased dose group are evaluator and subject-blinded. The increased frequency group is not blinded. Clinical assessments of disease activity will be based the European League Against Rheumatism (EULAR) criteria for response. Safety parameters will be assessed at every infusion.

A disease flare is defined by an increase in DAS28 with 0.6 or more at screening, when compared to the DAS28 score measured immediately prior to the last Remicade® infusion and depends upon the actual score as well. Since prior to enrollment, the subject received Remicade® as per routine clinical practice, the days on which infusions were administered and assessments are done during the induction period do not have to be exactly at Week 2, 6 and 14.

* Drug: Infliximab Control (double-blinded)
* Drug: Infliximab Increased Dose (double-blinded)
* Drug: Infliximab Increased Frequency (open-label)

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or more
* with RA according to ACR criteria
* presented with a disease flare after initial response to infliximab, with both response and flare being defined using the DAS28 score (EULAR criteria)
* received the standard Remicade® dosing schedule per the EU label (3 mg/kg at Weeks 0, 2, 6, [and 14])
* an initial response documented by moderate or good DAS28 improvement (EULAR criteria) from Week 0 to Week 6 or 14.

Exclusion Criteria:

* a female who is, or intends to become, pregnant during or within 6 months of the end of the study, is nursing or not using adequate contraceptive measures
* has not observed the designated periods for concomitant medications
* used any investigational medical product within 30 days prior to Baseline
* any clinically significant deviation from normal in the physical examination or chest X-ray that in the investigator's judgment, may interfere with the study evaluation or affect subject safety
* rheumatic disease other than RA or has any systemic inflammatory condition with signs and symptoms that might confound the evaluations of safety and toxicity
* allergic reaction/sensitivity to the study drug or its excipients that requires corticosteroid pre-infusion medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2006-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Increased Dose: 3 mg/kg infliximab + 1 extra vial (100 mg) infliximab every 8 weeks
Period: Overall Study
Arm/Group | Increased Dose | Increased Frequency | Control
Started | 14 | 11 | 18
Completed | 6 | 8 | 11
Not Completed | 8 | 3 | 7
Not completed — Adverse Event | 2 | 1 | 2
Not completed — Lack of Efficacy | 2 | 2 | 3
Not completed — Protocol Violation | 4 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Increased Dose | Increased Frequency | Control | Total
Number analyzed (Participants) | 14 | 11 | 18 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (13.0) | 58.6 (16.1) | 57.7 (12.3) | 58.3 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 14 | 34
  Male | 3 | 2 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in Disease Activity Score Based on 28 Joint Count (DAS28) Score.
Description: Descriptive summary of DAS28 (Disease Activity Score Based on 28 Joint Count)change from Baseline to the end of study (Week 24) in the population with available data at both Baseline and Week 24 (increased dose group, n=5; increased frequency group, n=7; and control group, n=5). DAS28 is a unit scale from 2.0 (best value) to 10.0 (worst value).
Time Frame: Between Screening (Week <=1) and Week 24
Population: Intent-to-treat population; subjects with available data at both Baseline and Week 24
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Increased Dose | Increased Frequency | Control
Number analyzed (Participants) | 5 | 7 | 5
Score on a Scale | -0.4 (1.27) | -1.6 (1.23) | -1.0 (1.90)

ADVERSE EVENTS:
Arm/Group | Infliximab*3mg/kg+1*Vial Q8W | Infliximab*3mg/kg Q6W | Control*Infliximab*3mg/kg Q8W
Serious Adverse Events (participants affected / at risk) | 2/14 | 0/11 | 2/18
Other Adverse Events (participants affected / at risk) | 7/14 | 5/11 | 5/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab*3mg/kg+1*Vial Q8W (N=14) | Infliximab*3mg/kg Q6W (N=11) | Control*Infliximab*3mg/kg Q8W (N=18)
VERTIGO (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
ASTHENIA (General disorders) | 0 (0) | 0 (0) | 1 (1)
INFUSION RELATED REACTION (General disorders) | 1 (1) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 1 (1)
ANAPHYLACTIC REACTION (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
BRAIN STEM SYNDROME (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
SOMNOLENCE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab*3mg/kg+1*Vial Q8W (N=14) | Infliximab*3mg/kg Q6W (N=11) | Control*Infliximab*3mg/kg Q8W (N=18)
ANAEMIA (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
CARDIOVASCULAR DISORDER (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
TINNITUS (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 1 (1) | 0 (0) | 0 (0)
LARYNGITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
PURULENT DISCHARGE (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
TINEA MANUUM (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
TOOTH INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
HEPATIC ENZYME INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
BURSITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
SUFFOCATION FEELING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0)
ANGIODYSPLASIA (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No